CLINICAL TRIAL: NCT04633356
Title: EUS Guided Portal-systemic Pressure Gradient Measurement in Patients With Chronic Hepatitis.
Brief Title: EUS Guided Portal-systemic Pressure Gradient Measurement
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Anthony Teoh, Associate Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017.519
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Portal Hypertension; Cirrhosis
Keywords: portal hypertension; portal pressure gradient; EUS interventions; Cirrhosis
MeSH Terms: conditions — Hypertension, Portal; Fibrosis

STUDY DESIGN:
Intervention Model Description: Patients recruited to the study would receive measurement of the portal pressure gradient with the use of the EUS-guided technique
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- EUS-portal pressure gradient measurement (PPGM) (Experimental): All patients would receive measurement of PPGM using the study device
  Interventions: Device: EUS-portal pressure gradient measurement (PPGM)

INTERVENTIONS:
Device: EUS-portal pressure gradient measurement (PPGM) — EUS-guided PPGM is performed under conscious sedation. An OGD would be performed to evaluate for findings consistent with portal hypertension such as varices and portal hypertensive gastropathy. The linear array echoendoscope is passed from the mouth into the stomach and duodenum, as with a standard exam. Under endoscopic ultrasound guidance, a 25 gauge EUS needle (Echotip, Cook Medical, USA) primed with heparin 100 USP/ml is then placed across the stomach or duodenal wall and through the liver parenchyma into the portal vein. A pressure measurement is then obtained from the compact pressure transducer attached to the handle of the needle. Three separate measurements are made with re-priming of heparin (less than 0.5 ml). The process is repeated for the hepatic vein. The EUS - PPG is calculated by subtracting the average of the three hepatic vein pressure measurements from the average of the 3 direct portal vein pressure measurements.

SUMMARY:
Portal hypertension is characterised by an increased portal pressure gradient (PPG), that is the difference in pressure between the portal vein and the inferior vena cava (IVC). Portal hypertension is a consequence of cirrhosis resulting from chronic hepatitis. Patients with portal hypertension are at risk of developing complications including oesophageal or gastric varices, variceal bleeding, ascites, spontaneous bacterial peritonitis, hepatic encephalopathy and mortality.

Albeit its clinical significance, direct measurement of portal venous pressure to document portal hypertension has traditionally been difficult. The portal vein pressure can be measured by transhepatic or transvenous methods but the procedure carries a risk of intra-peritoneal bleeding. Furthermore, the IVC pressure measurement requires further transjugular catheterisation. Hence, the technique is rarely used. Currently, the gold standard in measurement of portal hypertension is via measurement hepatic venous pressure gradient (HVPG). The HVPG has been shown to correlate with risk of clinical decompensation, development of varices, hepatocellular carcinoma, variceal bleeding, spontaneous bacterial peritonitis and mortality. Nevertheless, the technique has a low acceptance rate amongst patients and it may not be available even in tertiary medical centres.

Recently, the use of EUS-guided approach for measurement of portal pressure gradient (PPGM) has been shown to be feasible. The technical success rate was 100% and no adverse events were reported. Measurements obtained with the EUS approach was shown to correlate excellently with clinical parameters of portal hypertension including presence of varices, portal hypertensive gastropathy and thrombocytopenia. Furthermore, the procedure could be performed at the same time of screening oesophagogastroduodenoscopy (OGD), that is frequently required for variceal screening in this group of patients. Hence, the aim of the current study is to investigate the feasibility of EUS-PPGM and correlate the risk of developing complications with the PPGM in patients that are suffering from chronic hepatitis.

DETAILED DESCRIPTION:
Currently, the gold standard in measurement of portal hypertension is via measurement hepatic venous pressure gradient (HVPG). The HVPG has been shown to correlate with risk of clinical decompensation, development of varices, hepatocellular carcinoma, variceal bleeding, spontaneous bacterial peritonitis and mortality. The technique involves ultrasound guided puncture of the internal jugular vein, followed by passage of a balloon catheter from through the right atrium, IVC and right hepatic vein. The free hepatic vein venous pressure is then measured followed by the wedge balloon venous pressure. The HVPG is then calculated by subtracting the free hepatic venous pressure from the wedge balloon venous pressure. When HVPG is >10mmHg, the risk of developing varices is increased. If >12mmHg, then risk of variceal bleeding is increased. Mortality risk is increased when HVPG is >16-20mmHg. Nevertheless, the technique is technically difficult and it may not be available even in tertiary medical centres [8]. Furthermore, it requires the use of ionic contrast and also has a low acceptance rate amongst patients.

The aim of the current study is to investigate the feasibility of EUS-PPGM using the novel device and correlate the risk of developing complications with the PPGM in patients that are suffering from chronic hepatitis.

Recently, the use of EUS-guided approach for measurement of portal pressure gradient (PPGM) has been shown to be feasible. PPGM by the EUS approach was found to have excellent accuracy and strong correlation with pressure values obtained by the criterion standard transjugular wedged and free hepatic venous pressure measurements by interventional radiology in an animal model. Furthermore, in a pilot study involving 29 patients. The technical success rate was 100% and no adverse events were reported. Measurements obtained with the EUS approach was shown to correlate excellently with clinical parameters of portal hypertension including presence of varices, portal hypertensive gastropathy and thrombocytopenia. Furthermore, the procedure could be performed at the same time of screening oesophagogastroduodenoscopy (OGD), that is frequently required for variceal screening in this group of patients. However, whether the technique could reproduce results similar to HVPG in humans is uncertain.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from chronic hepatitis induced cirrhosis
* Informed consent available

Exclusion Criteria:

* Medical
* Child-Pugh Class C
* Uncorrected platelet count <50,000
* INR > 1.5 (natural)
* Anatomical
* Previous transjugular intrahepatic or surgical portosystemic shunt
* Portal vein thrombosis
* Anatomic alterations of the hepatic vasculature that prevent access to the portal vein or intrahepatic portion of the hepatic veins (identified at screening and/or during the endoscopic procedure).
* Previous history of spontaneous bacterial peritonitis within the previous three months
* Portopulmonary hypertension
* Cardiac decompensation
* Endoscopically Confirmed Exclusion Criteria
* Evidence of active GI bleeding (identified at screening and/or during the endoscopic procedure)
* If the volume of ascites in the path of the needle prevents apposition of the gastrointestinal tract and liver.
* Presence of gastric or duodenal ulcers, dieulafoy's lesion or cancers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-11-12 (Actual); Primary Completion 2024-11-11 (Estimated); Study Completion 2024-11-11 (Estimated)

PRIMARY OUTCOMES:
Technical success | 30 days
  Ability to place a needle in the portal and hepatic vein for calculation of portal pressure gradient

SECONDARY OUTCOMES:
Adverse events | 30 day
  Any untoward event directly arising from the measurement of PPGM

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang JY, Samarasena JB, Tsujino T, Lee J, Hu KQ, McLaren CE, Chen WP, Chang KJ. EUS-guided portal pressure gradient measurement with a simple novel device: a human pilot study. Gastrointest Endosc. 2017 May;85(5):996-1001. doi: 10.1016/j.gie.2016.09.026. Epub 2016 Sep 29. PMID 27693644
- [Background] Huang JY, Samarasena JB, Tsujino T, Chang KJ. EUS-guided portal pressure gradient measurement with a novel 25-gauge needle device versus standard transjugular approach: a comparison animal study. Gastrointest Endosc. 2016 Aug;84(2):358-62. doi: 10.1016/j.gie.2016.02.032. Epub 2016 Mar 3. PMID 26945557